CLINICAL TRIAL: NCT03971669
Title: Collection of Blood Samples for In-Vitro Studies from Healthy Adult Blood Donors Who Have Received Oral Typhoid Vaccine (TY21A)
Brief Title: Blood Donor CVD 5000
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Wilbur Chen, MD, MS, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00040022
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Risk Reduction
Keywords: Typhoid
MeSH Terms: conditions — Risk Reduction Behavior; Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Volunteers who choose to take part in this study will receive the licensed FDA-approved Oral Typhoid Vaccine (Vivotif).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccination with Oral Typhoid Vaccine (Vivotif) (Experimental): Volunteers receive immunization with Vivotif oral typhoid vaccine. Blood, saliva, and stool specimens are collected at subsequent visits.
  Interventions: Drug: Vivotif Typhoid Oral Vaccine

INTERVENTIONS:
Drug: Vivotif Typhoid Oral Vaccine — The 4 doses (1 capsule each) will be administered on alternate days, e.g., days 0, 2, 4, and 7 (± 1 day) under the supervision of the study coordinator(s).
  Other Names: Ty21a Typhoid Oral Vaccine

SUMMARY:
This is an open-label, non-randomized study. Volunteers will be vaccinated with the typhoid oral vaccine, Vivotif. Vivotif has been licensed by the Food and Drug Administration (FDA) for travelers to developing countries. Volunteers will also be asked to provide blood, saliva, and stool specimens over a follow-up time period of up to eight years. The specimens obtained in this clinical research study will be used to further the investigator's understanding of the protective immunological mechanisms that can be elicited systemically and may be applicable to other enteric pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Good general health as determined by a screening evaluation within 28 days before blood donation
* Informed, written consent

Exclusion Criteria:

* History of any of the following medical illnesses:

  * Diabetes
  * Cancer in past 5 years (except for basal cell carcinoma of the skin and cervical carcinoma in situ)
  * Heart disease (Hospitalization for a heart attack, coronary artery bypass graft, arrhythmia, or syncope, within past 5 years. Current symptoms of heart disease - dyspnea, angina, orthopnea)
  * Recurrent infections (more than 3 hospitalizations for invasive bacterial infections such as pneumonia or meningitis)
  * Current drug or alcohol abuse
  * Active ulcer disease or ongoing intestinal condition
  * Treatment for anemia in last 6 months
  * Currently being treated with anti-malarial drugs
* Any of the following laboratory abnormalities detected during medical screening:

  * WBC <0.81 x LLN or > 1.09 x ULN
  * Hemoglobin <0.91 x LLN or >1.18 x ULN (women) or <0.92 x LLN or >1.18 x ULN (men)
  * Platelet count <0.8 x LLN or > 1.2 x ULN
  * (For leukopheresis or blood unit donations, the following lab values are exclusionary:
  * WBC <3.5 or >11 x 103/mm3;
  * Hemoglobin <12.5 or >18 g/dl
  * Platelet count <150 or >500 x 103/mm3)
  * SGOT or SGPT >1.5 times normal
  * Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen
  * Positive serology for hepatitis B core antibody
  * Poor peripheral venous access for blood donation
  * Positive RPR
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or interfere with the scientific integrity of study.
* Positive urine pregnancy test (HCG) on day of vaccination. Prior to each blood donation -females with menstrual history consistent with pregnancy. Pregnant women will not be enrolled, because immunological changes that occur during pregnancy may interfere with laboratory assays.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-01-16 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders | approximately 5 years
  Percentage of responders by cytokine production (Interferon-gamma (IFN-gamma) or Tumor Necrosis Factor-alpha (TNF-α)) by mass cytometry or flow cytometry. Responders will be defined as those volunteers showing increases post-immunization of >0.1% of positive CD8+ cells for IFN-gamma or TNF-α over baseline (pre-immunization) values.) or Tumor Necrosis Factor-alpha (TNF-α)) by mass cytometry or flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States